CLINICAL TRIAL: NCT00368069
Title: A Double-blind, Placebo-controlled, Randomized Efficacy and Safety Study of Keppra® Extended Release Formulation - XR Once Daily as add-on Therapy in Subjects From 12 to 70 Years With Refractory Epilepsy Suffering From Partial Onset Seizures.
Brief Title: A Study to Look at the Efficacy and Safety of Keppra® Extended Release Formulation - XR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01235; 2006-000987-10 (EudraCT Number)
Record Dates: First submitted 2006-08-11; First posted 2006-08-24 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Keppra® XR; Levetiracetam XR; Extended release
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Keppra® XR (Experimental): Keppra® extended release formulation -XR
  Interventions: Drug: Keppra® extended release formulation - XR
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Keppra® extended release formulation - XR — 500mg extended release oral tablet, 2 tablets once daily
  Other Names: Levetiracetam XR
  Arms: Keppra® XR
Drug: Placebo — oral tablets, 2 tablets once daily
  Arms: Placebo

SUMMARY:
This is a safety and efficacy study of Keppra® extended release formulation - XR in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of refractory epilepsy
* Patients must be receiving a stable dose of 1 - 3 concomitant Anti-Epileptic Drugs (AED)
* Female patients without childbearing potential. Female patients with childbearing potential are eligible if they use a medically accepted non-hormonal contraceptive method

Exclusion Criteria:

* Seizures occurring in clusters
* Status epilepticus within 3 months of Visit 1
* History of non-epileptic seizures
* Known allergic reaction or intolerance to pyrrolidine derivatives and/or excipients
* Pregnant or lactating women. Any woman with childbearing potential who is not using a medically accepted, non-hormonal method of birth control

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2006-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (34):
- N01235 1007, Curitiba, Brazil
- Finland (3):
  - N01235 2001, Kuopio
  - N01235 2003, Tampere
  - N01235 2002, Turku
- India (10):
  - N01235 3008, Chennai
  - N01235 3010, Chennai
  - N01235 3012, Gandhinagar
  - N01235 3003, Hyderabad
  - N01235 3004, Hyderabad
  - N01235 3001, Lucknow
  - N01235 3009, Madurai
  - N01235 3002, Mumbai
  - N01235 3007, Mumbai
  - N01235 3011, Visakhapatnam
- Mexico (4):
  - N01235 4006, Aguascalientes
  - N01235 4003, Distrio Federal
  - N01235 4001, Guadalajara
  - N01235 4005, Puebla City
- Russia (9):
  - N01235 5001, Moscow
  - N01235 5002, Moscow
  - N01235 5003, Moscow
  - N01235 5005, Moscow
  - N01235 5006, Moscow
  - N01235 5007, Moscow
  - N01235 5004, Saint Petersburg
  - N01235 5009, Saint Petersburg
  - N01235 5008, Smolensk
- South Africa (2):
  - N01235 6002, Cape Town
  - N01235 6003, Umhlanga
- Ukraine (5):
  - N01235 7001, Kharkiv
  - N01235 7004, Kharkiv
  - N01235 7005, Lviv
  - N01235 7002, Odesa
  - N01235 7003, Poltava

REFERENCES:
- [Result] Peltola J, Coetzee C, Jimenez F, Litovchenko T, Ramaratnam S, Zaslavaskiy L, Lu ZS, Sykes DM; Levetiracetam XR N01235 Study Group. Once-daily extended-release levetiracetam as adjunctive treatment of partial-onset seizures in patients with epilepsy: a double-blind, randomized, placebo-controlled trial. Epilepsia. 2009 Mar;50(3):406-14. doi: 10.1111/j.1528-1167.2008.01817.x. PMID 19317886
- [Result] Richy FF, Banerjee S, Brabant Y, Helmers S. Levetiracetam extended release and levetiracetam immediate release as adjunctive treatment for partial-onset seizures: an indirect comparison of treatment-emergent adverse events using meta-analytic techniques. Epilepsy Behav. 2009 Oct;16(2):240-5. doi: 10.1016/j.yebeh.2009.07.013. Epub 2009 Aug 20. PMID 19699156
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The N01235 study began recruitment in August 2006 with study completion occurring in May 2007.
Pre-assignment Details: Baseline and Participant Flow data consists of the Intent-to-Treat (ITT) analysis group. The ITT group consists of all randomized subjects.
Groups:
- Keppra®: Keppra® extended release formulation (XR)
Period: Overall Study
Arm/Group | Keppra® | Placebo
Started | 79 | 79
Completed | 71 | 72
Not Completed | 8 | 7
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal of Consent | 2 | 1
Not completed — no blood sampling possible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Keppra® | Placebo | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.97 (13.41) | 32.38 (12.60) | 33.17 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 59
  Male | 52 | 47 | 99
Region of Enrollment [Number; unit: participants]
  Mexico | 15 | 16 | 31.0
  Finland | 2 | 2 | 4.0
  Ukraine | 13 | 12 | 25.0
  South Africa | 4 | 4 | 8.0
  Russian Federation | 19 | 19 | 38.0
  India | 25 | 26 | 51.0
  Brazil | 1 | 0 | 1.0

OUTCOME MEASURES:

1. Primary Outcome: Partial Onset Seizure (POS) Frequency Per Week - Intention-To-Treat (ITT) Population
Description: Number of POS over the treatment period standardized to 1 week period.
Time Frame: Treatment period (12 weeks)
Population: Intention-to-treat (ITT) (Analyses were performed on subjects from the ITT with non-missing information during baseline and treatment period.)
Measure: Least Squares Mean (Standard Error); unit: seizures per week (log-transformed data)
Arm/Group | Keppra® | Placebo
Number analyzed (Participants) | 75 | 78
seizures per week (log-transformed data) | 0.912 (0.053) | 1.067 (0.052)
Statistical Analysis 1: Comparison: Keppra® vs Placebo; Test type: Superiority or Other; p = 0.038, ANCOVA; Analysis of covariance (ANCOVA) on (log-) POS freq/week over Treatment period with Treatment, (log-) Baseline POS freq/week as covariate; Mean Difference (Net) = 0.155, 95% CI [0.009 to 0.301]
Statistical Analysis 2: Comparison: Keppra® vs Placebo; Treatment difference was assessed through the percent reduction in POS freq/week of Keppra over Placebo by back transformation of the results of the ANCOVA on log data; Test type: Superiority or Other; Transf. of ANCOVA results on log data; Percent Reduction of Keppra over PBO is calculated based on the ANCOVA on log data as 100*(1-exp(LSmeans Keppra -LSMeans Placebo)); Percent reduction over Placebo = 14.4, 95% CI [0.9 to 26.0]

2. Secondary Outcome: POS Seizure Frequency Per Week Over Baseline and Treatment Period
Time Frame: Baseline Period (8 weeks) - Treatment Period (12 weeks)
Population: ITT Population - no imputation techniques used for missing data (number of subjects with non-missing data for Baseline = ITT Population and for Treatment period = 75 patients for levetiracetam and 78 patients for PBO) Clusters of type I count are included in the count of Type I seizures
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Keppra® | Placebo
Number analyzed (Participants) | 79 | 79
seizures per week
  Baseline POS frequency per week | 1.80 [1.13 to 4.13] | 2.11 [1.33 to 3.26]
  Treatment POS frequency per week | 0.99 [0.33 to 2.70] | 1.36 [0.92 to 2.85]

3. Secondary Outcome: All (Type I+II+III) Seizures Frequency Per Week
Description: Number of All type Seizures over the treatment period standardized to 1 week period (Type I -Partial Onset Seizures, Type II - Generalized Seizures, Type III - Unclassified Epileptic Seizures)
Time Frame: Treatment period (12 weeks)
Population: ITT (Analyses were performed on subjects from the ITT with non-missing information during baseline and treatment period.)
Measure: Least Squares Mean (Standard Error); unit: seizures per week (log-transformed data)
Arm/Group | Keppra® | Placebo
Number analyzed (Participants) | 75 | 78
seizures per week (log-transformed data) | 0.928 (0.053) | 1.086 (0.052)
Statistical Analysis 1: Comparison: Keppra® vs Placebo; Test type: Superiority or Other; p = 0.034, ANCOVA; ANCOVA on (log-) seizure frequency per week over Treatment period with Treatment, (log-) Baseline seizure frequency per week as covariate; Mean Difference (Net) = 0.158, 95% CI [0.012 to 0.305]
Statistical Analysis 2: Comparison: Keppra® vs Placebo; Treatment difference was assessed through the percent reduction in POS frequency per week of Keppra over Placebo by back transformation of the results of the ANCOVA on log data; Test type: Superiority or Other; Transf. of ANCOVA results on log data; Percent Reduction of Keppra over Placebo is calculated based on the ANCOVA on log data as 100*(1-exp(LSmeans Keppra -LSMeans Placebo)); Percent reduction over Placebo = 14.7, 95% CI [1.2 to 26.3]

4. Secondary Outcome: 50% Response in Weekly POS Frequency
Description: A subject is considered as a 50% responder in POS if he/she has a >= 50% decrease from Baseline in the POS frequency/week over Treatment period.
Time Frame: Treatment period (12 weeks)
Population: ITT Based on the number of evaluable patients. A patient is considered as evaluable for the response status if he has seizure information in at least one of the periods (baseline or treatment period)
Measure: Number; unit: Participants
Arm/Group | Keppra® | Placebo
Number analyzed (Participants) | 79 | 79
Participants
  Response | 34 | 23
  Non-Response | 45 | 56
Statistical Analysis 1: Comparison: Keppra® vs Placebo; Test type: Superiority or Other; p = 0.070, Regression, Logistic; Logistic regression analysis including Treatment as a factor; Odds Ratio (OR) = 1.84, 95% CI [0.95 to 3.55] — Based on the number of evaluable patients. A patient is considered as evaluable for the response status if he has seizure information in at least one of the period (baseline or treatment period

5. Secondary Outcome: Response in Weekly POS Frequency (Categorized Into 6 Categories According to Reduction) Over the Treatment Period of 12 Weeks
Description: The response is classified according to the percent reduction from baseline in the POS frequency per week over the Treatment Period of 12 weeks duration.
Time Frame: over the treatment period (12 weeks)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Keppra® | Placebo
Number analyzed (Participants) | 79 | 79
Participants
  < -25% | 11 | 13
  -25% - <25% | 14 | 23
  25% - <75% | 35 | 34
  75% - <100% | 11 | 7
  100% | 8 | 2
Statistical Analysis 1: Comparison: Keppra® vs Placebo; Test type: Superiority or Other; p = 0.033, Mantel Haenszel; Subjects with missing data during the Treatment period were considered in the category <-25%

6. Primary Outcome: Partial Onset Seizure (POS) Frequency Per Week - Per Protocol (PP) Population
Description: Number of POS over the treatment period standardized to 1 week period
Time Frame: Treatment Period (12 weeks)
Population: Per Protocol (PP) Population (Analyses were performed on subjects from the PP Population with non-missing information during both baseline and treatment period)
Measure: Least Squares Mean (Standard Error); unit: seizures per week (log-transformed data)
Arm/Group | Keppra® | Placebo
Number analyzed (Participants) | 67 | 69
seizures per week (log-transformed data) | 0.914 (0.049) | 1.119 (0.048)
Statistical Analysis 1: Comparison: Keppra® vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA on (log-) Treatment POS frequency per week with Treatment and (log-) Baseline POS frequency per week as covariate; Mean Difference (Net) = 0.205, 95% CI [0.070 to 0.341]
Statistical Analysis 2: Comparison: Keppra® vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; Transf. of ANCOVA results on log data; [statistical method as in outcome 3, analysis 2]; Percent reduction over Placebo = 18.6, 95% CI [6.7 to 28.9]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Selection Visit (Week 0) until Final Visit (Week 22).
Description: Adverse Event reporting is data is taken from the Safety Set (SS) analysis group. The SS is comprised all subjects who were dispensed study medication.
Arm/Group | Keppra® | Placebo
Serious Adverse Events (participants affected / at risk) | 6/77 | 2/79
Other Adverse Events (participants affected / at risk) | 23/77 | 21/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keppra® (N=77) | Placebo (N=79)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keppra® (N=77) | Placebo (N=79)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Irritability (General disorders) | 5 (5) | 0 (0)
Influenza (Infections and infestations) | 6 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 5 (6) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 5 (8) | 11 (21)
Somnolence (Nervous system disorders) | 6 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.